CLINICAL TRIAL: NCT04468607
Title: A Phase I, Open-Label, Dose-Escalation Study Of The Safety And Pharmacokinetics Of BLYG8824A Administered Intravenously In Patients With Locally Advanced Or Metastatic Colorectal Cancer
Brief Title: A Study of BLYG8824A in Participants With Locally Advanced or Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GO41751; 2023-503409-12-00 (EU CTIS Number)
Record Dates: First submitted 2020-06-23; First posted 2020-07-13 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose-Escalation Stage (Experimental): Participants will be assigned sequentially to escalating doses of BLYG8824A, up to the maximum tolerated dose (MTD).
  Interventions: Drug: BLYG8824A
- Dose-Expansion Stage (Experimental): Once dose escalation is completed and the MTD (or MAD) has been identified, a recommended expansion dose will be proposed for the dose-expansion stage of the trial.
  Interventions: Drug: BLYG8824A

INTERVENTIONS:
Drug: BLYG8824A — BLYG8824A will be administered at a flat dose independent of body weight.
  Other Names: linclatamig; RG6286

SUMMARY:
This study will evaluate the safety, tolerability, and pharmacokinetics of BLYG8824A and will make a preliminary assessment of the anti-tumor activity of BLYG8824A in patients with locally advanced or metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status of 0 or 1
* Life expectancy of at least 12 weeks
* Histologically or cytologically documented invasive CRC: incurable, unresectable, locally advanced or metastatic CRC previously treated with multimodality therapy or mCRC
* Locally advanced or metastatic CRC that has relapsed or is refractory to established therapies
* Prior disease progression (or intolerance) following oxaliplatin, irinotecan, fluoropyrimidines, and anti-EGFR monoclonal antibodies
* An archival tissue specimen or fresh baseline biopsy (when archival is not available) is required for enrollment into the study
* Measurable disease, according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Non-measurable evaluable disease is acceptable for dose-escalation.
* Adequate hematologic and end organ function
* Acute, clinically significant treatment-related toxicity from prior therapy resolved to Grade ≤ 1 prior to study entry

Expansion Cohort-Specific Inclusion Criteria

* MSS or MSI-L disease as determined by polymerase chain reaction (PCR) and/or IHC
* Measurable disease by RECIST v1.1 with at least one measurable target lesion in the expansion cohort
* Progression must have occurred during or after most recent treatment for locally advanced or metastatic colorectal cancer
* For patients enrolled in either a dedicated biopsy cohort or other expansion cohorts where biopsy is clinically feasible, willingness to consent to mandatory fresh pretreatment and on-treatment biopsies of safely accessible tumor lesions

Exclusion Criteria:

* Pregnant or breastfeeding, or intending to become pregnant during the study or within 4 months after the final dose of BLYG8824A
* Significant cardiopulmonary dysfunction
* Known clinically significant liver disease
* Positive serologic or PCR test results for acute or chronic HBV infection
* Acute or chronic HCV infection
* HIV seropositivity
* Poorly controlled Type 2 diabetes mellitus
* Current treatment with medications that are well known to prolong the QT interval
* Primary CNS malignancy, untreated CNS metastases, or active CNS metastases
* Leptomeningeal disease
* Spinal cord compression that has not been definitively treated with surgery and/or radiation
* History of autoimmune disease
* Prior allogeneic stem cell or solid organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2024-10-16 (Actual)

PRIMARY OUTCOMES:
Incidence and Nature of DLTs | Approximately 48 months
Number of Patricipants with Adverse Events | Approximately 48 months
Number Of Cycles Received | Approximately 48 months
Dose Intensity | Approximately 48 months
Maximum Tolerated Dose(s) MTD(s) of BLYG8824A | Approximately 48 months

SECONDARY OUTCOMES:
Serum Concentration of BLYG8824A | At predifined interevals from Cycle 1 Day 1; Cycle 2 Day 1; Cycles ≥ 3, Day 1; Treatment Completion/ Discontinuation (Cycle length: 21 days)
Overall Response Rate (ORR) | Approximately 48 months
  ORR is defined as the proportion of patients with a complete response (CR) or partial response (PR) as determined by the investigator according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1)
Duration of Response (DOR) | Approximately 48 months
  Duration of response (DOR), defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause (whichever occurs first), as determined by the investigator according to RECIST v1.1
Presence of Anti-drug Antibodies (ADAs) | Cycle 1, Day 1; Cycle 2 Day 1; Cycles ≥ 3, Day 1; Treatment Completion/ Discontinuation (Cycle length: 21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (6):
- United States (2):
  - City of Hope, Duarte, California
  - SCRI Oncology Partners, Nashville, Tennessee
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia
- Spain (3):
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - START Madrid-FJD, Hospital Fundacion Jimenez Diaz, Madrid

IPD SHARING:
Plan to Share IPD: No